CLINICAL TRIAL: NCT06757140
Title: Opioid Drug Interactions: Safety, Abuse Potential and Pharmacokinetic Effects
Brief Title: Opioid Drug Interaction Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanna Babalonis, PhD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Shanna Babalonis, PhD, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 97946; R01DA016718 (NIH)
Record Dates: First submitted 2024-12-09; First posted 2025-01-03 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Drug Interactions; Drug Kinetics
Keywords: inpatient study; opioids; opiates; sedatives; opioid misuse
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Alprazolam; Oxycodone; oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Placebo / Placebo (Placebo Comparator): Participants will receive 2 drug administrations, neither will be active. The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for both alprazolam and oxycodone ≈ 1.5 hr).
  Interventions: Drug: Placebo
- Placebo / Oxycodone low oral dose (Percocet, Roxicodone) (Experimental): Participants will receive 2 drug administrations, one dose oral placebo and one low dose oral oxycodone. The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for both alprazolam and oxycodone ≈ 1.5 hr).
  Interventions: Drug: Oxycodone; Drug: Placebo
- Placebo / Oxycodone high oral dose (Percocet, Roxicodone) (Experimental): Participants will receive 2 drug administrations, one dose oral placebo and one high dose oral oxycodone. The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for both alprazolam and oxycodone ≈ 1.5 hr).
  Interventions: Drug: Oxycodone; Drug: Placebo
- Alprazolam low oral dose (Xanax) / Placebo (Experimental): Participants will receive 2 drug administrations, one dose oral placebo and one low dose oral alprazolam. The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for both alprazolam and oxycodone ≈ 1.5 hr).
  Interventions: Drug: Alprazolam; Drug: Placebo
- Alprazolam high oral dose (Xanax) / Placebo (Experimental): Participants will receive 2 drug administrations, one dose oral placebo and one high dose oral alprazolam. The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for both alprazolam and oxycodone ≈ 1.5 hr).
  Interventions: Drug: Alprazolam; Drug: Placebo
- Alprazolam low oral dose (Xanax) / Oxycodone low oral dose (Percocet, Roxicodone) (Experimental): Participants will receive 2 non-therapeutic oral drug administrations, one low dose alprazolam, and one low dose oxycodone. The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for both alprazolam and oxycodone ≈ 1.5 hr).
  Interventions: Drug: Alprazolam; Drug: Oxycodone
- Alprazolam high oral dose (Xanax) / Oxycodone low oral dose (Percocet, Roxicodone) (Experimental): Participants will receive 2 non-therapeutic oral drug administrations, one high dose alprazolam, and one low dose oxycodone. The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for both alprazolam and oxycodone ≈ 1.5 hr).
  Interventions: Drug: Alprazolam; Drug: Oxycodone
- Alprazolam low oral dose (Xanax) / Oxycodone high oral dose (Percocet, Roxicodone) (Experimental): Participants will receive 2 non-therapeutic oral drug administrations, one low dose alprazolam, and one high dose oxycodone. The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for both alprazolam and oxycodone ≈ 1.5 hr).
  Interventions: Drug: Alprazolam; Drug: Oxycodone
- Alprazolam high oral dose (Xanax) / Oxycodone high oral dose (Percocet, Roxicodone) (Experimental): Participants will receive 2 non-therapeutic oral drug administrations, one high dose alprazolam, and one high dose oxycodone. The experimental sessions are designed to capture the time-action curves for the test drugs (Tmax for both alprazolam and oxycodone ≈ 1.5 hr).
  Interventions: Drug: Alprazolam; Drug: Oxycodone

INTERVENTIONS:
Drug: Alprazolam — Participants will receive varying non-therapeutic experimental doses of oral alprazolam, alone and in combination with oral oxycodone
  Other Names: Xanax
  Arms: Alprazolam high oral dose (Xanax) / Oxycodone high oral dose (Percocet, Roxicodone); Alprazolam high oral dose (Xanax) / Oxycodone low oral dose (Percocet, Roxicodone); Alprazolam high oral dose (Xanax) / Placebo; Alprazolam low oral dose (Xanax) / Oxycodone high oral dose (Percocet, Roxicodone); Alprazolam low oral dose (Xanax) / Oxycodone low oral dose (Percocet, Roxicodone); Alprazolam low oral dose (Xanax) / Placebo
Drug: Oxycodone — Participants will receive varying non-therapeutic experimental doses of oral oxycodone, alone and in combination with oral alprazolam
  Other Names: Percocet; Roxicodone
  Arms: Alprazolam high oral dose (Xanax) / Oxycodone high oral dose (Percocet, Roxicodone); Alprazolam high oral dose (Xanax) / Oxycodone low oral dose (Percocet, Roxicodone); Alprazolam low oral dose (Xanax) / Oxycodone high oral dose (Percocet, Roxicodone); Alprazolam low oral dose (Xanax) / Oxycodone low oral dose (Percocet, Roxicodone); Placebo / Oxycodone high oral dose (Percocet, Roxicodone); Placebo / Oxycodone low oral dose (Percocet, Roxicodone)
Drug: Placebo — Participants will receive inactive oral doses
  Arms: Alprazolam high oral dose (Xanax) / Placebo; Alprazolam low oral dose (Xanax) / Placebo; Placebo / Oxycodone high oral dose (Percocet, Roxicodone); Placebo / Oxycodone low oral dose (Percocet, Roxicodone); Placebo / Placebo

SUMMARY:
This study will examine the effects of doses of opioid/placebo and doses of alprazolam/placebo, alone and in combination. The primary outcomes are pharmacodynamic measures (subjective ratings of drug liking and other abuse-related effects; physiological outcomes) and pharmacokinetic outcomes (from blood samples) to determine the interaction effects of these compounds.

DETAILED DESCRIPTION:
Alprazolam (Xanax®) is a short-acting benzodiazepine that is the commonly prescribed in the U.S. (>15 million prescriptions in 2021) and CDC reporting indicates that alprazolam was associated with the greatest increase in number of ED presentations of the benzodiazepines. This study will examine the effects of a widely prescribed and abused mu opioid agonist, oxycodone, and a widely prescribed and abused benzodiazepine, alprazolam, when given alone and in combination to experienced drug using volunteers. Key safety outcomes, including expired CO2, pharmacodynamic measures related to abuse potential, and cognitive/psychomotor performance will be thoroughly examined over a range of doses for both drugs alone and in combination. Pharmacokinetic data will also be collected and analyzed to assess the potential pharmacokinetic interaction as an underlying mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking and literate participants, able to understand and sign Informed Consent Document
* ages 18 to 55 years old inclusive
* BMI of greater than/equal to 17 and approximately less than or equal to 30
* self-reported opioid use
* self-reported sedative-like drug use
* women of childbearing potential must not be pregnant or breastfeeding at screening and be using an effective form of contraception throughout study participation
* otherwise healthy as determined by the medical/research team based on medical history, physical examination, vital signs, laboratory chemistries (blood chemistry with liver function tests and hematology, urinalysis and microscopic evaluation, 12-lead electrocardiogram)
* willing and able to comply with all testing requirements defined in the protocol
* adequate venous access (determined by RN) for pharmacokinetic blood draws

Exclusion Criteria:

* physical dependence on alcohol, opioids, benzodiazepines or sedative/hypnotics requiring medical management/detoxification
* seeking treatment for opioid or any other drug use
* acute medical problem (e.g., infection) or chronic medical problem requiring daily medication or ongoing medical care (e.g., hypertension, cardiovascular disease, diabetes, respiratory disorders [e.g., asthma, COPD])
* clinically significant abnormal ECG (as determined by study physician/cardiologist)
* clinically significant abnormal laboratory findings (e.g., liver function tests greater than 3x the upper limits of normal range)
* current or past history of major psychiatric disorder that would limit ability to participate in the study (e.g., bipolar disorder).
* recent use of CYP2C9, CYP2D6 and CYP3A4 inhibitor or inducer that is long-acting and not amenable to a wash-out period after enrollment
* known hypersensitivity to any of the study drugs
* currently pregnant or breastfeeding
* currently under parole or probation with urine testing requirements

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Subject-Rated Outcome: Visual Analog Scale (VAS) Drug Liking | This outcome was recorded prior to and in regular intervals after drug administration for the duration of the session (approx. 6.5 hours per session).
  Participants rated their subjective drug liking on a standardized VAS scale (0 to 100) with higher scores equating to increased liking. Raw data transformed to peak scores.

SECONDARY OUTCOMES:
Change in Subject-Rated Outcome: Visual Analog Scale (VAS) Drug Effect | This outcome was recorded prior to and in regular intervals after drug administration for the duration of the session (approx. 6.5 hours per session).
  Participants rated their subjective drug effect on a standardized VAS scale (0 to 100) with higher scores equating to increased effect. Raw data transformed to peak scores.
Change in Respiration Rate | Respiration rate recorded prior to and in regular intervals after drug administration for the duration of the session (approx. 6.5 hours per session).
  Respiration rate monitored throughout each session. Raw data transformed to trough scores.
Change in End-tidal Carbon Dioxide (EtCO2) | End-tidal Carbon Dioxide (EtCO2) recorded prior to and in regular intervals after drug administration for the duration of the session (approx. 6.5 hours per session).
  Change in End-tidal Carbon Dioxide (EtCO2) monitored throughout each session. Raw data transformed to peak scores.
Change in Oxygen Saturation | Oxygen Saturation recorded prior to and in regular intervals after drug administration for the duration of the session (approx. 6.5 hours per session).
  Oxygen Saturation monitored throughout each session. Raw data transformed to trough scores.

CONTACTS AND LOCATIONS:
Overall Officials: Shanna Babalonis, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP